CLINICAL TRIAL: NCT01470105
Title: Improving a Bayesian Model's Survival Estimates in Patients Needing Surgery for Bone Metastases
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 11-121
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Bone Metastases
Keywords: questionnaire; 11-121
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood

GROUPS / COHORTS (1):
- pts bone metastases: This is a prospective, cross sectional, human use study conducted using patients with bone metastases requiring orthopaedic stabilization. Though this is an observational study, blood sampling, the SF-36 questionnaire, and ECOG performance status, and correlative studies will be performed.
  Interventions: Other: blood sampling, the SF-36 questionnaire

INTERVENTIONS:
Other: blood sampling, the SF-36 questionnaire — The patient be asked to fill out a questionnaire. The questionnaire asks about their quality of life and will take approximately 15 minutes to complete. It will be completed at a regularly scheduled clinic visit.
  At the scheduled pre-operative testing, an extra sample of your blood (equal to about 4 teaspoons) will be collected for research tests. The research tests will measure levels of inflammation in your body. These tests are not part of routine care. A physical examination of the operative site will be done by the Orthopaedic Surgeon. The patient will complete the same questionnaire at the regularly scheduled three and six month follow-up visit

SUMMARY:
The goal of this study is to improve how we estimate survival of people with cancer that has spread to their bone. There have been previous attempts to estimate survival of people with cancer that spread to the bone, but they have not been accurate. This study will try to improve the way we estimate survival in people with cancer that has spread to their bone by looking to see if a physician assessment and a patient assessment of the health status can be blended to give a better estimate of survival than patients or doctors alone.

ELIGIBILITY:
Inclusion Criteria:

* ≥ to 18 years of age
* Diagnosed with a metastatic malignancy
* histologically proven in oligometastatic disease or by clinical suspicion in widely metastatic disease
* by conventional radiographs, cross sectional imaging and/or scintigraphy
* Scheduled for an orthopaedic operative intervention for skeletal metastases at MSKCC or Montefiore Medical Center including, not limited to the following:
* Resection
* Intramedullary Fixation
* Prophylactic fixation
* Curettage and cementation
* Internal fixation
* Arthroplasty
* Spine stabilization

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential subjects will be recruited by the Orthopaedic Service of the Department of Surgery.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2011-11; Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
serum inflammatory cytokines | 3 years
  Whether the addition of serum inflammatory cytokines improves the robustness of an existing, validated Bayesian Belief network trained to estimate survival in human patients with operative skeletal metastases.

SECONDARY OUTCOMES:
chemokine analysis | 3 years
  Whether the addition of chemokine analysis improves the robustness of an existing, validated Bayesian Belief network trained to estimate survival in human patients with operative skeletal metastases.
patient-reported SF-36 data | 3 years
  Whether the addition of and inclusion of patient-reported SF-36 data, improves the robustness of an existing, validated Bayesian Belief network trained to estimate survival in human patients with operative skeletal metastases.

CONTACTS AND LOCATIONS:
Overall Officials: Carol Morris, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm